CLINICAL TRIAL: NCT03519295
Title: A Non-comparative Randomized 2:1 Phase II Study of Docetaxel, Cisplatin, and 5-fluorouracil in Combination or Not With Atezolizumab in Patients With Metastatic or Unresectable Locally Advanced Squamous Cell Anal Carcinoma
Brief Title: A Study of mDCF in Combination or Not With Atezolizumab in Advanced Squamous Cell Anal Carcinoma
Acronym: SCARCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCARCE C17-02
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Anal Cancer
Keywords: Epidermoid Cancers of the Anal Canal
MeSH Terms: conditions — Anus Neoplasms | interventions — atezolizumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A - mDCF + Atezolizumab (Experimental): * MPDL3280A (atezolizumab) will be administered every 2 weeks at 800 mg for 12 months.
  * Patients will receive 8 cycles of mDCF (docetaxel 40 mg/m2 day 1, cisplatin 40 mg/m2 day 1 and 5FU at 1200 mg/m2/day for 2 days) every 2 weeks
  Interventions: Drug: MPDL3280A; Drug: mDCF
- ARM B - mDCF (Active Comparator): Patients will receive 8 cycles of mDCF (docetaxel 40 mg/m2 day 1, cisplatin 40 mg/m2 day 1 and 5FU at 1200 mg/m2/day for 2 days) every 2 weeks.
  Interventions: Drug: mDCF

INTERVENTIONS:
Drug: MPDL3280A — MPDL3280A administered every 2 weeks at 800 mg for 12 months.
  Other Names: atezolizumab
  Arms: ARM A - mDCF + Atezolizumab
Drug: mDCF — 8 cycles of mDCF (docetaxel 40 mg/m2 day 1, cisplatin 40 mg/m2 day 1 and 5-FU at 1200 mg/m2/day for 2 days) every 2 weeks
  Other Names: modified docetaxel, cisplatin, and fluorouracil

SUMMARY:
SCARCE is a non-comparative randomized, 2:1 phase II study. The purpose of this study is to assess the progression-free survival rate at 12 months. (evaluation according with RECISTv1.1 criteria).

For all patients, CT scan will be planned at baseline, and every 8 weeks until 12 months from randomization (or disease progression), and every 12 weeks thereafter.

PET scan will be performed at baseline, at the end of mDCF treatment, and at 12 months after randomization (in absence of disease progression).

CT scan and PET scan will be collected for a centralized review.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the anal canal (SCCA) is a rare disease, its incidence increases worldwide and no standard therapy is currently available to treat metastatic or relapsing cases. SCCA is mostly induced by human papillomavirus (HPV) infections with HPV-related oncoproteins (E6 and E7) expressed in more than 90% of cases.

Based on the preliminary results of the Epitope-HPV02 study and although it provide proof of concept data on taxane-based chemotherapy efficacy in SCCA, complete responses observed after 6-8 cycles of chemotherapy has not translated into long-term remissions .

Combining immunogenic chemotherapy with anti-PD-1/PD-L1 might be a convenient way to increase the diversity of antigens released by tumor and T cells.

So for the SCARCE study, we hypothesized that combination of mDCF (8 cycles) with MPDL32801 (12 months) might induce synergy and improve the rate of long-term PFS rate.

The aim of the SCARCE study is to provide a valuable proof of concept to establish immunogenic chemotherapy and anti-PDL1 as a standard of care for SCCA patients with poor clinical outcomes and to take advantage of the presence of HPV antigens in most patients (HPV 16 and 18 genotypes are involved in 90% of SCCA) to set up a specific immunomonitoring program based on tumor samples and blood-derived lymphocytes to better understand the potential synergisms between immunogenic chemotherapy and anti-PDL1 and to identify valuable biomarkers of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years,
2. Performance status Eastern Cooperative Oncology Group World Health Organization (ECOG-WHO) ≤1,
3. Histologically proven and unresectable locally advanced recurrent or metastatic squamous cell anal carcinoma,
4. Presence of a target lesion on CT-scan assessed by RECIST v1.1 criteria,
5. Patient eligible to the mDCF regimen,
6. CT scan performed within 28 days prior inclusion,
7. PET scan performed within 28 days prior inclusion,
8. Signed and dated informed consent,
9. Patient affiliated to or beneficiary of French social security system,
10. Ability to comply with the study protocol, in the Investigator's judgment,
11. Life expectancy ≥ 6 months,
12. Adequate hematologic and end-organ function.
13. Previous concomitant chemoradiotherapy is permitted if completed before 28 days of starting treatment.

Exclusion Criteria:

Non-eligibility to clinical trials if one of the following parameter is reported:

1. Previously received chemotherapy for metastatic disease,
2. Previously received cisplatin except for concomitant chemoradiotherapy,
3. Previously received taxanes (paclitaxel or docetaxel) or another spindle poison (navelbine) in the treatment of SCCA,
4. Previously received anti-tumor immunotherapy (HPV vaccination is allowed),
5. Previous radiotherapy within 28 days of randomization (14 days if radiotherapy of bone metastases)
6. Diagnosis of additional malignancy within 3 years prior to the randomization with the exception for curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical or breast cancer,
7. Any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study,
8. Current participation in a study of an investigational agent or in the period of exclusion,
9. Pregnancy, breast-feeding or absence/refusal of adequate contraception for fertile patients during the period of treatment and for 6 months from the last treatment administration, men must refrain from donating sperm during this same period.
10. Patient under guardianship, curatorship or under the protection of justice.

    Non-eligible to chemotherapy:
11. Inadequate organ functions: uncontrolled cardiac condition, known cardiac failure, unstable coronaropathy, respiratory failure, and Chronic Obstructive Pulmonary Disease (COPD),
12. Diabetes with vascular or neurovascular complications,
13. Preexistent peripheral neuropathy or impaired audition,
14. HIV positive with CD4 count under 400 cells/mm3 (VIH test is mandatory before inclusion),
15. Active hepatitis B or C virus (HBV or HCV) infection (chronic or acute), (Defined as having a positive HBV surface antigen (HBsAg) test at screening. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total HBV core antibody (HBcAb) test at screening, are eligible for the study. HCV infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test),
16. Active tuberculosis,
17. Concomitant treatment with CYP3A4 inhibitor like ritonavir, indinavir, or ketoconazole, etc. Replacement by another drug before randomization, whenever is possible, is allowed,
18. Known hypersensitivity or contraindication to any of the study chemotherapy drugs (taxanes, cisplatin, 5FU), according with the SmPC of each drug
19. Uncontrolled infection or another life-risk condition,
20. Known hearing impairment that contraindicates cisplatin administration,
21. Administration of a live (attenuated) vaccine within 28 days of planned start of study therapy of known need for this vaccine during treatment,
22. Administration of prophylactic phenytoin,
23. Inadequate laboratory values: creatinine clearance (CrCl by Modification of Diet in Renal Disease [MDRD] formula) <60 ml/min, neutrophil count <1500 /mm3, platelets <100000/mm3, bilirubin 2.5 x upper limit of normal (ULN), aspartate transaminase (AST)/alanine transaminase (ALT) 2.5 x ULN or 5 x ULN with liver metastasis.
24. Patient with known dihydropyridine dehydrogenase (DPD) deficiency or history of severe and unexpected reactions to a fluoropyrimidine-containing regimen, or in case of clinically significant active heart disease or myocardial infarction within 6 months or if patient treated with sorivudine or its clinically related analogues, such as brivudine

    Non-eligible to immunotherapy:
25. Any immunosuppressive therapy (i.e. corticosteroids >10mg of hydrocortisone or equivalent dose) within 14 days before the planned start of study therapy,
26. Active autoimmune disease that has required a systemic treatment in past 2 years (i.e. corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin) is allowed.

    Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, (see Annex 7 for a more comprehensive list of autoimmune diseases and immune deficiencies) with the following exceptions:
27. Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study,
28. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study,
29. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area,
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids,
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months,
30. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
31. Known active central nervous system metastases and/or carcinomatous meningitis. Subject with previously treated brain metastases and with radiological and clinical stability are allowed,
32. Previously received an anti-PD1, anti-PDL1, or anti-CTLA4 agent,
33. Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of atezolizumab formulation,
34. History of colorectal inflammatory disease,
35. History of idiopathic or secondary pulmonary fibrosis (history of radiation pneumonitis in the radiation field fibrosis is permitted), or evidence of active pneumonitis requiring a systemic treatment with 28 days before the planned start of study therapy,
36. Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study,
37. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia,
38. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate (PFS) | at 12 months
  PFS will be defined as the time interval between the date of randomization and the date of first progression (local, regional, metastatic, second cancer) or death regardless of the cause. Patients alive without progression will be censored at the time of the latest news

SECONDARY OUTCOMES:
Overall Survival (OS) | within 3 years after the initiation of the treatment
  OS will be calculated between the date of randomization and the date of death from any cause. . Alive patients or lost to follow-up at the time of the analysis will be censored at the date of last follow-up.
Progression free survival | within 3 years after the initiation of the treatment
  PFS will be defined as the time interval between the date of randomization and the date of first progression (local, regional, metastatic, second cancer) or death regardless of the cause
Quality of life related to heath | From the randomization to patient death or for maximum 3 years
  EORTC-QLQ-C30
Objective response rate (ORR) | within 3 years after the initiation of the treatment
  Evaluated by RECIST criteria version 1.1
Tolerance graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] criteria v4.03 | within 3 years after the initiation of the treatment
  graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] criteria v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Stefano KIM, MD, Principal Investigator — University Hospital of Besançon
Locations (31):
- France (31):
  - Clinique de l'Europe, Amiens
  - Institut Sainte Catherine, Avignon
  - CHRU Jean Minjoz, Besançon
  - CHU Bordeaux - Hôpital Haut Lévêque, Bordeaux
  - Centre François Baclesse, Caen
  - Hôpitaux Civils de Colmar, Colmar
  - Clinique des Cèdres, Cornebarrieu
  - GHPSO Creil, Creil
  - Centre Georges François Leclerc, Dijon
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Oscar Lambert, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Jean Mermoz, Lyon
  - CHU Timone, Marseille
  - Hopital Montbéliard, Montbéliard
  - ICM Val d'Aurelle, Montpellier
  - CHU Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Antoine, Paris
  - Groupe Hospitalier Diaconesses Crois Saint Simon, Paris
  - Groupe Hospitalier Saint Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Henri Mondor, Paris
  - Hôpital saint Louis, Paris
  - Insitut Curie, Paris
  - Centre CARIO, Plérin
  - CHU Poitiers, Poitiers
  - CHU Robert Debré Reims, Reims
  - CH Saint Quentin, Saint-Quentin
  - Centre Paul Strauss, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim S, Ghiringhelli F, de la Fouchardiere C, Evesque L, Smith D, Badet N, Samalin E, Lopez-Trabada Ataz D, Parzy A, Desrame J, Baba Hamed N, Buecher B, Tougeron D, Bouche O, Dahan L, Chibaudel B, El Hajbi F, Mineur L, Dubreuil O, Ben Abdelghani M, Pecout S, Bibeau F, Herfs M, Garcia ML, Meurisse A, Vernerey D, Taieb J, Borg C. Atezolizumab plus modified docetaxel, cisplatin, and fluorouracil as first-line treatment for advanced anal cancer (SCARCE C17-02 PRODIGE 60): a randomised, non-comparative, phase 2 study. Lancet Oncol. 2024 Apr;25(4):518-528. doi: 10.1016/S1470-2045(24)00081-0. PMID 38547895
- [Derived] Kim S, Buecher B, Andre T, Jary M, Bidard FC, Ghiringhelli F, Francois E, Taieb J, Smith D, de la Fouchardiere C, Desrame J, Samalin E, Parzy A, Baba-Hamed N, Bouche O, Tougeron D, Dahan L, El Hajbi F, Jacquin M, Rebucci-Peixoto M, Spehner L, Vendrely V, Vernerey D, Borg C. Atezolizumab plus modified docetaxel-cisplatin-5-fluorouracil (mDCF) regimen versus mDCF in patients with metastatic or unresectable locally advanced recurrent anal squamous cell carcinoma: a randomized, non-comparative phase II SCARCE GERCOR trial. BMC Cancer. 2020 Apr 25;20(1):352. doi: 10.1186/s12885-020-06841-1. PMID 32334548